CLINICAL TRIAL: NCT01535430
Title: Assessment of Reorganization and Plasticity of Eloquent Function in Patients With Brain Tumors
Brief Title: Assessment of Eloquent Function in Brain Tumor Patients
Status: Recruiting | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0240-24-FB; 0671-11-FB (Other: UNMC original paper protocol #)
Record Dates: First submitted 2012-02-08; First posted 2012-02-17 (Estimated); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Primary Brain Tumor; Metastatic Brain Tumor
Keywords: brain mapping; brain tumor
MeSH Terms: conditions — Brain Neoplasms | interventions — Brain Mapping

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Eloquent area tumor: Standard of care with brain mapping, pre-, intra-, and post-operative.
  Interventions: Diagnostic Test: Brain mapping

INTERVENTIONS:
Diagnostic Test: Brain mapping — Brain mapping will be employed pre-, intra-, and post-operatively to evaluate specific functions.

SUMMARY:
Purpose of the study:

AIM 1: Prospectively collect pre-operative [functional magnetic resonance imaging (fMRI), diffusion tensor imaging (DTI), magnetoencephalography (MEG)] and intra-operative mapping data in patients with intra-axial brain tumors to assess how well each modality predicts the location of eloquent brain function. In addition, each modality will be compared with the other.

AIM 2: Assess reorganization of eloquent brain function and plasticity in patients with intra-axial brain tumors. This will be accomplished by prospectively collecting post-operative mapping studies and neuropsychological tests to compare them to prior mapping studies as stated above.

DETAILED DESCRIPTION:
Any patient with a primary or metastatic brain tumor in or near an eloquent area would be eligible for participation in the study assuming no contraindications to any of the studies or operative procedure.

Pre-operative evaluation will include clinical evaluation, neuropsychological testing, magnetic resonance imaging (MRI) brain with and without contrast, fMRI, DTI tractograms, and MEG studies as well as standard pre-operative work-up.

Intra-operative procedures include all non-invasive pre-operative mapping data being incorporated into the operative procedure with imaging tools that are routinely used during neurosurgical procedures. Participants will have awake mapping performed. Usual standards of care will be followed during craniotomy, mapping, and tumor resection or biopsy.

Post-operative procedures include routine post-operative care and assessment consisting of clinical examinations and imaging obtained within 24 hours post-resection. Participants will have routine follow-up outpatient appointments after surgery which will include neurologic assessment and follow-up imaging (MRI with and without contrast) for their tumors as appropriate. The experimental portion of the protocol is incorporating repeat neuropsychological testing and mapping studies (fMRI, DTI, MEG) studies at 2 and 6 months post-surgery into their routine follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 19 years and older
* Brain tumor in or near eloquent brain regions that is appropriate for attempted resection
* Appropriate body habitus and mental status/capacity to participate with non-invasive or invasive mapping
* Benign or malignant intra-axial brain tumor
* Primary or metastatic intra-axial brain tumor

Exclusion Criteria:

* Any contraindication to MRI (i.e. implanted devices)
* Inappropriate body habitus or mental status/capacity to participate with non-invasive or invasive mapping in a safe and reliable manner
* Declining to participate
* Lacks capacity to understand the study or consent for themselves
* Neurologic status which precludes testing (poor function- not testable)
* Positive pregnancy test
* End stage renal disease or severe renal dysfunction

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with a brain tumor in or near an area of eloquent brain function (speech, motor, sensory).
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2012-01-31 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Eloquent function | 1 year
  The location of the eloquent function of interest (motor, sensory, speech) will be assessed pre-operatively and intra-operatively and compared. Then, at 2 and 6 months post-operatively, repeat non-invasive mapping studies will be performed to compare to the subjects' prior studies. This will allow for assessment of reorganization and plasticity of function. Additionally, novel ways of identifying eloquent brain regions will be developed.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Aizenberg, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ellis DG, White ML, Hayasaka S, Warren DE, Wilson TW, Aizenberg MR. Accuracy analysis of fMRI and MEG activations determined by intraoperative mapping. Neurosurg Focus. 2020 Feb 1;48(2):E13. doi: 10.3171/2019.11.FOCUS19784. PMID 32006951